CLINICAL TRIAL: NCT05442554
Title: A Phase 4, Single Arm, Open Label, Multicenter Study of Brentuximab Vedotin Treatment of Chinese Patients With CD30-Positive Cutaneous T-Cell Lymphoma
Brief Title: A Study of Brentuximab Vedotin Treatment in Chinese Adults With CD30-Positive Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C25029
Record Dates: First submitted 2022-06-30; First posted 2022-07-05 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: T-Cell Lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brentuximab Vedotin (Experimental): Participants received brentuximab vedotin 1.8 milligrams per kilogram (mg/kg), IV on Day 1 of each 21-day cycle for up to a total of 16 cycles.
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin — Brentuximab vedotin IV infusion.
  Other Names: SGN-35

SUMMARY:
The main aim is to check the long-term side effects of treatment with Brentuximab Vedotin and to see if that treatment improves symptoms of cluster of differentiation antigen 30 (CD30-Positive) Cutaneous T-Cell Lymphoma in Chinese adults.

Participants will receive brentuximab vedotin through the vein on day 1 of each 21 day cycle up to maximum 16 cycles.

DETAILED DESCRIPTION:
The drug being tested in this study is called brentuximab vedotin (SGN-35). Brentuximab vedotin is being tested to treat people who have CD30-positive cutaneous T-Cell lymphoma.

The study will enroll approximately 10 patients. Participants will receive a single treatment i.e., brentuximab vedotin monotherapy:

• Brentuximab vedotin 1.8 mg/kg

Participants will be administered with brentuximab vedotin by intravenous (IV) infusion given for approximately 30 minutes on Day 1 of each 21-day cycle up to 16 cycles followed by the end of treatment (EOT) visit 30 days after receiving the final dose of study drug. Participants with progressive disease (PD) at any time during the study will be discontinued from study drug.

This multi-center trial will be conducted in China. Participants will remain in this study for approximately 56 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically- confirmed cluster of differentiation antigen 30 positive (CD30+) disease by local laboratory assessment and pathology review.

2. Participants with primary cutaneous anaplastic large cell lymphoma (pcALCL) who have received prior radiation therapy or at least 1 prior systemic therapy, or participants with mycosis fungoides (MF) who have received at least 1 prior systemic therapy for their disease. 3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2. 4. Suitable venous access for the study-required blood sampling. 5. Participants must have radiographically or clinically measurable or evaluable disease.

6. Recovered (i.e., Grade 1 toxicity) from the reversible effects of prior antineoplastic therapy.

-Exclusion Criteria:

1. A concurrent diagnosis of systemic anaplastic large cell lymphoma (ALCL), or other non-Hodgkin lymphoma (excluding lymphomatoid papulosis [LyP]).
2. A concurrent diagnosis of sézary syndrome (SS) or high blood tumor burden (B2) disease.
3. Corticosteroid therapy for the treatment of cutaneous T-cell lymphoma (CTCL) within 3 weeks of first dose of study drug.
4. Known hypersensitivity to recombinant proteins, murine proteins, or any excipient contained in the drug formulation.
5. Life-threatening illness unrelated to cancer.
6. Severe central nervous system (CNS), pulmonary, renal, or hepatic disease not related to the participant's cancer.
7. Known active cerebral/meningeal disease, including signs or symptoms of progressive multifocal leukoencephalopathy (PML).
8. Known human immunodeficiency virus (HIV) positive.
9. Known hepatitis B surface antigen positive or known or suspected active hepatitis C infection.
10. Any severe active systemic viral, bacterial, or fungal infection within 1 week before first study drug dose requiring systemic antimicrobial therapy. (Oral antibiotics for prophylaxis are allowed.)
11. Receiving antibody-directed or immunoglobulin-based immune therapy (eg, immunoglobulin replacement, other monoclonal antibody therapies) within 12 weeks of first study drug dose.
12. Any of the following cardiovascular conditions or values within 6 months before the first dose of study drug:

    * Myocardial infarction within 6 months of enrollment.
    * New York Heart Association (NYHA) Class III or IV heart failure.
    * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
13. History of another primary malignancy not in remission for at least 3 years. The following are exempt from the 3-year limit: completely resected in situ carcinoma, such as nonmelanoma skin cancer and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Pap smear.
14. Oral retinoid therapy for any indication within 3 weeks of the first dose of study drug.
15. History of pancreatitis or significant risk factors for developing pancreatitis (eg, prior pancreatitis, uncontrolled hyperlipidemia, excessive alcohol consumption, uncontrolled diabetes mellitus, biliary tract disease, and medications known to increase triglyceride levels or to be associated with pancreatic toxicity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (4):
- China (4):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
Takeda does not provide access to Individual Participant Data when a study is in a very limited (small) study population due to participant privacy concerns such as potential reidentification of study participants.

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/52b934f938554c0e?idFilter=%5B%22VedolizumabSC-4003%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in China from 28 November 2022 to 09 August 2024.
Pre-assignment Details: Participants with cluster of differentiation 30-positive mycosis fungoides (CD30+ MF) or primary cutaneous anaplastic large cell lymphoma (pcALCL) histologically confirmed by local pathology assessment participated in the study to receive brentuximab vedotin.
Groups:
- Brentuximab Vedotin: Participants received brentuximab vedotin 1.8 milligrams per kilogram (mg/kg), intravenously (IV) on Day 1 of each 21-day cycle for up to a total of 16 cycles.
Period: Overall Study
Arm/Group | Brentuximab Vedotin
Started | 10
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all enrolled participants who received at least 1 dose of study drug.
Groups:
- Brentuximab Vedotin: Participants received brentuximab vedotin 1.8 mg/kg, IV on Day 1 of each 21-day cycle for up to a total of 16 cycles.
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Lasting at Least 4 Months in Participants With CD30+ MF or pcALCL
Description: ORR is defined as the percentage of participants who achieve complete response (CR) or partial response (PR) that lasts at least 4 months. CR is defined as complete disappearance of all clinical evidence of disease and PR is defined as regression of measurable disease. ORR was determined based on Global Response Score (GRS) which consisted of a skin assessment by the investigator using the modified severity-weighted assessment tool (mSWAT), nodal and visceral involvement using computed tomography (CT) scan, and for the participants with mycosis fungoides (MF) only, detection of circulating Sezary cells. Response Criteria were based on International Society for Cutaneous Lymphomas (ISCL), United States Cutaneous Lymphoma Consortium (USCLC) and European Organisation for Research and Treatment of Cancer (EORTC) Consensus guidelines.
Time Frame: Up to 58 weeks
Population: The response-evaluable population included a subset of the full analysis set (FAS) participants with measurable disease at baseline and with at least 1 post-baseline response assessment. FAS consisted of all enrolled participants identified as CD30+ and received at least 1 dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
percentage of participants | 60.0 [26.2 to 87.8]

2. Secondary Outcome: Complete Response (CR) Rate
Description: CR rate is defined as the percentage of participants with CR. CR is defined as complete disappearance of all clinical evidence of disease. CR was determined based on GRS which consisted of a skin assessment by the investigator using the mSWAT, nodal and visceral involvement using computed tomography (CT) scan, and for the participants with MF only, detection of circulating Sezary cells. Response Criteria were based on ISCL, USCLC and EORTC Consensus guidelines.
Time Frame: Up to 58 weeks
Population: The response-evaluable population included a subset of the FAS participants with measurable disease at baseline and with at least 1 post-baseline response assessment. FAS consisted of all enrolled participants identified as CD30+ and received at least 1 dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
percentage of participants | 0 [0 to 30.8]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve complete response (CR) or partial response (PR). CR is defined as complete disappearance of all clinical evidence of disease and PR is defined as regression of measurable disease. ORR was determined based on GRS which consisted of a skin assessment by the investigator using the mSWAT, nodal and visceral involvement using CT scan, and for the participants with MF only, detection of circulating Sezary cells. Response Criteria were based on ISCL, USCLC and EORTC Consensus guidelines.
Time Frame: Up to 58 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
percentage of participants | 70.0 [34.8 to 93.3]

4. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was assessed in participants with CR or PR and is defined as the time between first documentation of response and progressive disease (PD). Response criteria were based on ISCL, USCLC and EORTC Consensus guidelines. Participants who were lost to follow-up, withdrew consent, or discontinued treatment due to undocumented PD after the last adequate disease assessment were censored at the last disease assessment.
Time Frame: Up to 58 weeks
Population: The response-evaluable population included a subset of the FAS participants with measurable disease at baseline and with at least 1 post-baseline response assessment. FAS consisted of all enrolled participants identified as CD30+ and received at least 1 dose of the study drug. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 7
months | NA [NA to NA] — Median and confidence interval (CI) was not estimable as no participants with the event were reported.

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g. a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. TEAE is defined as an adverse event with an onset that occurs after receiving study drug. SAE is any AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event. TEAE and SAE were determined as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (up to approximately 58 weeks)
Population: The safety analysis set consisted of all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
Participants
  TEAEs | 10
  SAEs | 4

6. Secondary Outcome: Changes From Baseline in Participant's Vital Sign: Systolic and Diastolic Blood Pressure
Description: Vital signs included seated blood pressure (systolic and diastolic) measurements.
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: The safety analysis set consisted of all enrolled participants who received at least 1 dose of study drug. Number of participants analyzed is the number of participants with data available for analysis at the specified time points.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
millimeters of mercury (mmHg)
  Systolic Blood Pressure: Baseline | 125.6 (11.04)
  Systolic Blood Pressure: Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Systolic Blood Pressure: Change from Baseline at the End of Treatment | -2.9 (8.81)
  Diastolic Blood Pressure: Baseline | 76.5 (6.36)
  Diastolic Blood Pressure: Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Diastolic Blood Pressure: Change from Baseline at the End of Treatment | -4.4 (4.61)

7. Secondary Outcome: Changes From Baseline in Participant's Vital Sign: Heart Rate
Description: Vital signs included heart rate (beats per minute) measurements.
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
beats per minute
  Baseline | 87.4 (10.11)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Change from Baseline at the End of Treatment | -10.3 (14.34)

8. Secondary Outcome: Changes From Baseline in Participant's Vital Sign: Body Temperature
Description: Vital signs included body temperature (degree Celsius) measurements.
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: degree Celsius (°C)
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
degree Celsius (°C)
  Baseline | 36.62 (0.368)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Change from Baseline at the End of Treatment | 0.00 (0.361)

9. Secondary Outcome: Number of Participants From Baseline to Worst Post-Baseline Assessment Categories Based on Eastern Cooperative Oncology Group (ECOG) Performance Status Scale
Description: ECOG scale was used to assess performance status of participants. Grades range from 0 (fully active) to 5 (dead) where Grade 0: Normal activity. Grade 1: Symptoms but ambulatory. Grade 2: In bed <50% of the time. Grade 3: In bed >50% of the time. Grade 4: 100% bedridden. Grade 5: Dead. Lower grades indicate improvement. Reported here is the number of participants in each reported baseline grade to their worst post-baseline grade assessment on the ECOG scale.
Time Frame: Baseline up to 30 days after the last dose of study drug (up to approximately 58 weeks)
Population: The safety analysis set consisted of all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
Participants
  Participants with Baseline Grade: 0 to Worst Post-Baseline Grade: 0 | 2
  Participants with Baseline Grade: 1 to Worst Post-Baseline Grade: 1 | 7
  Participants with Baseline Grade: 1 to Worst Post-Baseline Grade: 3 | 1

10. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
grams per liter (g/L)
  Baseline | 126.3 (23.00)
  Change from baseline at the End of Treatment: number analyzed (Participants) | 9
  Change from baseline at the End of Treatment | -5.4 (16.46)

11. Secondary Outcome: Change From Baseline in Hematology Parameter: Neutrophil Count
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter (L)
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
10^9 cells/liter (L)
  Baseline | 3.949 (2.2230)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Change from Baseline at the End of Treatment | 0.189 (4.4084)

12. Secondary Outcome: Change From Baseline in Hematology Parameter: Platelet Count
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
10^9 cells/L
  Baseline | 279.2 (78.24)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Change from Baseline at the End of Treatment | -97.0 (86.87)

13. Secondary Outcome: Change From Baseline in Hematology Parameter: Lymphocyte Count
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
10^9 cells/L
  Baseline | 1.530 (0.7367)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Change from Baseline at the End of Treatment | -0.101 (0.3355)

14. Secondary Outcome: Change From Baseline in Hematology Parameter: Leukocyte Count
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
10^9 cells/L
  Baseline | 7.082 (3.1018)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Change from Baseline at the End of Treatment | -0.862 (3.5380)

15. Secondary Outcome: Change From Baseline in Serum Chemistry Parameter: Alkaline Phosphatase (ALP)
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
Units per liter (U/L)
  Baseline | 89.0 (29.66)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Change from Baseline at the End of Treatment | 26.3 (36.10)

16. Secondary Outcome: Change From Baseline in Serum Chemistry Parameter: Alanine Aminotransferase (ALT)
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
U/L
  Baseline | 18.9 (10.45)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Change from Baseline at the End of Treatment | 8.2 (15.52)

17. Secondary Outcome: Change From Baseline in Serum Chemistry Parameter: Aspartate Aminotransferase (AST)
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
U/L
  Baseline | 19.0 (5.85)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Change from Baseline at the End of Treatment | 10.7 (10.40)

18. Secondary Outcome: Change From Baseline in Serum Chemistry Parameter: Total Bilirubin
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: micromoles per liter (µmol/L)
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
micromoles per liter (µmol/L)
  Baseline | 8.82 (3.879)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 9
  Change from Baseline at the End of Treatment | 1.93 (3.947)

19. Secondary Outcome: Change From Baseline in Serum Chemistry Parameter: Lipase
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
U/L
  Baseline: number analyzed (Participants) | 8
  Baseline | 35.96 (10.726)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 7
  Change from Baseline at the End of Treatment | 4.90 (11.837)

20. Secondary Outcome: Change From Baseline in Serum Chemistry Parameter: Amylase
Time Frame: Baseline, at end of treatment (approximately Week 54)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
U/L
  Baseline: number analyzed (Participants) | 8
  Baseline | 64.0 (24.55)
  Change from Baseline at the End of Treatment: number analyzed (Participants) | 7
  Change from Baseline at the End of Treatment | 10.9 (25.80)

ADVERSE EVENTS:
Time Frame: Up to 58 weeks
Description: The safety analysis set consisted of all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Brentuximab Vedotin
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=10)
Dysuria (Renal and urinary disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Oedema peripheral (General disorders) | 1
Renal tubular necrosis (Renal and urinary disorders) | 1
White blood cell count decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=10)
Alanine aminotransferase increased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Amylase increased (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Aspartate aminotransferase increased (Investigations) | 2
Bile acids increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 2
Blood creatinine decreased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Constipation (Gastrointestinal disorders) | 1
Cystatin C increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 3
Gamma-glutamyltransferase increased (Investigations) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 2
Neutrophil count decreased (Investigations) | 2
Oedema peripheral (General disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Paraesthesia (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pyrexia (General disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 2
Red blood cell sedimentation rate increased (Investigations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tricuspid valve incompetence (Cardiac disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 2
White blood cell count increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT05442554/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT05442554/SAP_001.pdf